CLINICAL TRIAL: NCT04877483
Title: To Evaluate the Short-term and Long Term Efficacy of Acupuncture in Ocular and Oral Dryness Symptoms of Dry Eye Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-07-003C
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye Syndrome; Xerophthalmia
Keywords: dry eye syndromes; Xerophthalmia; acupuncture; GB20; BL2; Oral microbiota
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia | interventions — Acupuncture Therapy; Microbiota; Blood Cell Count

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group GB20 (Experimental): Group GB20 will received acupuncture at acupoint GB20 twice a week 8 weeks for efficacy evaluation. And we could use the oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Procedure: Acupuncture; Diagnostic Test: Oral microbiota; Diagnostic Test: Schirmer's test; Diagnostic Test: Tear breakup time; Diagnostic Test: OSDI(Ocular Surface Disease Index); Diagnostic Test: TCM pattern; Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: TCM pulse diagnosis; Diagnostic Test: TCM heart rate variability; Diagnostic Test: ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index); Diagnostic Test: Whole-genome genotyping(TWBv2.0); Diagnostic Test: Cytokine markers; Diagnostic Test: Blood biochemical analysis; Diagnostic Test: complete blood count (CBC); Diagnostic Test: SF-36(36-Item Short Form Survey )
- Group GB20 plus BL2 (Experimental): Group GB20 plus BL2 will received acupuncture at acupoint GB20 plus BL2 twice a week 8 weeks for efficacy evaluation. And we could use the oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Procedure: Acupuncture; Diagnostic Test: Oral microbiota; Diagnostic Test: Schirmer's test; Diagnostic Test: Tear breakup time; Diagnostic Test: OSDI(Ocular Surface Disease Index); Diagnostic Test: TCM pattern; Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: TCM pulse diagnosis; Diagnostic Test: TCM heart rate variability; Diagnostic Test: ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index); Diagnostic Test: Whole-genome genotyping(TWBv2.0); Diagnostic Test: Cytokine markers; Diagnostic Test: Blood biochemical analysis; Diagnostic Test: complete blood count (CBC); Diagnostic Test: SF-36(36-Item Short Form Survey )
- Healthy control (Other): Healthy control group will not received any treatment. And we could use the oral microbiota, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability to find the difference with the comparison between the dry eye syndrome and healthy control.
  Interventions: Diagnostic Test: Oral microbiota; Diagnostic Test: TCM pattern; Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: TCM pulse diagnosis; Diagnostic Test: TCM heart rate variability; Diagnostic Test: Whole-genome genotyping(TWBv2.0); Diagnostic Test: Cytokine markers
- Waiting list (Other): Group Waiting list will not received any treatment. at acupoint GB20 plus BL2 twice a week 8 weeks for efficacy evaluation. And we could use the oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Diagnostic Test: Oral microbiota; Diagnostic Test: Schirmer's test; Diagnostic Test: Tear breakup time; Diagnostic Test: OSDI(Ocular Surface Disease Index); Diagnostic Test: TCM pattern; Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: TCM pulse diagnosis; Diagnostic Test: TCM heart rate variability; Diagnostic Test: ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index); Diagnostic Test: Whole-genome genotyping(TWBv2.0); Diagnostic Test: Cytokine markers; Diagnostic Test: Blood biochemical analysis; Diagnostic Test: complete blood count (CBC); Diagnostic Test: SF-36(36-Item Short Form Survey )

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture is a form of treatment that inserting very thin needles through a person's skin at specific points on the body. Group GB20 and Group GB20 plus BL2 will received the acupuncture treatment.
  Arms: Group GB20; Group GB20 plus BL2
Diagnostic Test: Oral microbiota — Group GB20, Group GB20 plus BL2 and Healthy control will take the oral microbiota analysis.
Diagnostic Test: Schirmer's test — Group GB20 and Group GB20 plus BL2 will take the Schirmer's test.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: Tear breakup time — Group GB20 and Group GB20 plus BL2 will take the tear breakup time test.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: OSDI(Ocular Surface Disease Index) — Group GB20 and Group GB20 plus BL2 will take the OSDI test.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: TCM pattern — Group GB20, Group GB20 plus BL2 and Healthy control will take the Traditional Chinese Medicine pattern diagnosis.
Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis — Group GB20, Group GB20 plus BL2 and Healthy control will take the Traditional Chinese Medicine(TCM) tongue diagnosis.
Diagnostic Test: TCM pulse diagnosis — Group GB20, Group GB20 plus BL2 and Healthy control will take the Traditional Chinese Medicine(TCM) pulse diagnosis.
Diagnostic Test: TCM heart rate variability — Group GB20, Group GB20 plus BL2 and Healthy control will take the TCM Heart rate variability.
Diagnostic Test: ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index) — Group GB20 and Group GB20 plus BL2 will take the ESSPRI.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: Whole-genome genotyping(TWBv2.0) — Group GB20, Group GB20 plus BL2 and Healthy control will take the Whole-genome genotyping(TWBv2.0).
Diagnostic Test: Cytokine markers — Group GB20, Group GB20 plus BL2 and Healthy control will take the cytokine markers(IL-17、MMP-9、BAFF、BCMA) analysis.
Diagnostic Test: Blood biochemical analysis — Group GB20 and Group GB20 plus BL2 will take the Blood biochemical analysis(BUN,Cre,AST,ALT,ESR and CRP).
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: complete blood count (CBC) — Group GB20 and Group GB20 plus BL2 will take the CBC(WBC、RBC、Hb、Platelet) analysis.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list
Diagnostic Test: SF-36(36-Item Short Form Survey ) — Group GB20 and Group GB20 plus BL2 will take the SF-36 test.
  Arms: Group GB20; Group GB20 plus BL2; Waiting list

SUMMARY:
This study wants to use a randomized, single-blind, controlled trial to evaluate the efficacy of receiving acupuncture GB20 or GB20 plus BL2 on alleviating the ocular dryness symptom from dry eye syndrome and Sjögren's syndrome. One hundred dry eye syndrome subjects are composed of 50 dry eye syndrome subjects and 50 Sjögren's syndrome' dry eye subjects, and all are randomized into 40 Group GB20 and 40 Group GB20 plus BL2 (GBL), and 20 Group Waiting list; while we also include 20 healthy controls. Fifty dry eye syndrome subjects are randomized into 20 Group GB20, 20 Group GBL and 10 Group Waiting list in first year; while both Group GB20 or GBL received acupuncture twice a week 8 weeks for efficacy evaluation, and 10 Group Waiting list receive no any acupuncture treatment. And we could use the Whole-genome genotyping, oral microbiota, Schirmer's test, Tear breakup time, Cytokines, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose. In second year, another 50 dry eye syndrome subjects are also enrolled and randomized into randomized into 20 Group GB20, 20 Group GBL and 10 Group Waiting list; while both Group GB20 or GBL received acupuncture twice a week 8 weeks for efficacy evaluation with above outcome measurements, and 10 Group Waiting list receive no any acupuncture treatment. Meanwhile, we also include 20 healthy controls, and we want to find the difference with the comparison between the dry eye syndrome, Sjögren's syndrome and healthy control in second year. Through the analysis for dry eye syndrome and Sjögren's syndrome, we could find the biomarker to differentiate dry eye syndrome, Sjögren's syndrome and healthy control. In the future, this work could be applied for screening and diagnosis of pre-dry eye syndrome and Sjögren's syndrome, and this integrated TCM with Western Medicine plan could be applied for the goal of holistic health care.

DETAILED DESCRIPTION:
Method: This study wants to use a randomized, single-blind, controlled trial to evaluate the efficacy of receiving acupuncture GB20 or GB20 plus BL2 on alleviating the ocular dryness symptom from dry eye syndrome and Sjögren's syndrome. One hundred dry eye syndrome subjects are composed of 50 dry eye syndrome subjects and 50 Sjögren's syndrome' dry eye subjects, and all are randomized into 40 Group GB20 and 40 Group GB20 plus BL2 (GBL), and 20 Group Waiting list; while we also include 20 healthy controls. Fifty dry eye syndrome subjects are randomized into 20 Group GB20, 20 Group GBL and 10 Group Waiting list in first year; while both Group GB20 or GBL received acupuncture twice a week 8 weeks for efficacy evaluation, and 10 Group Waiting list receive no any acupuncture treatment. And we could use the Whole-genome genotyping, oral microbiota, Schirmer's test, Tear breakup time, Cytokines, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose. In second year, another 50 dry eye syndrome subjects are also enrolled and randomized into randomized into 20 Group GB20, 20 Group GBL and 10 Group Waiting list; while both Group GB20 or GBL received acupuncture twice a week 8 weeks for efficacy evaluation with above outcome measurements, and 10 Group Waiting list receive no any acupuncture treatment. Meanwhile, we also include 20 healthy controls, and we want to find the difference with the comparison between the dry eye syndrome, Sjögren's syndrome and healthy control in second year. Through the analysis for dry eye syndrome and Sjögren's syndrome, we could find the biomarker to differentiate dry eye syndrome, Sjögren's syndrome and healthy control. In the future, this work could be applied for screening and diagnosis of pre-dry eye syndrome and Sjögren's syndrome, and this integrated TCM with Western Medicine plan could be applied for the goal of holistic health care.

Expected Results:

1. To evaluate the difference among Schirmer's test, TBUT, TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis, heart rate variability, Whole-genome genotyping, oral microbiota, and Cytokines for dry eye syndrome, Sjögren's syndrome and healthy control.
2. Integrated functional multi-omics for dry eye syndrome and healthy control.
3. To evaluate the efficacy of GB20 plus BL2 for dry eye syndrome and Sjögren's syndrome.
4. To evaluate the efficacy of GB20 for dry eye syndrome and Sjögren's syndrome.
5. To evaluate the efficacy of BL2 for dry eye syndrome and Sjögren's syndrome.

Keywords: Dry eye syndrome, Sjögren's syndrome, Xerophthalmia, Acupuncture, GB20, BL2

ELIGIBILITY:
* Dry eye syndrome

  * Inclusion Criteria:

    1. aged between 20 and 75 years
    2. Schirmer's test less than 10 mm/5 min
  * Exclusion Criteria:

    1. Pregnancy
    2. With eye inflammation or infectious eye disease
    3. Accepted operation of eye
* Sjögren's syndrome

  * Inclusion Criteria:

    1. primary or secondary SS
    2. aged between 20 and 75 years
    3. fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
    4. had no abnormal findings of immune, liver, kidney, or blood function evaluations.
  * Exclusion Criteria:

    1. a history of alcohol abuse, diabetes mellitus, or major life-threatening condition
    2. pregnancy or breastfeeding
    3. steroid pulse therapy within three months prior to the commencement of our study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Schirmer's test | one year
  Schirmer's test is a tool for evaluating aqueous tear production among the dry eye syndrome.
OSDI(Ocular Surface Disease Index) | one year
  OSDI(Ocular Surface Disease Index) is a tool to rate the severity of dry eye disease among the dry eye syndrome.

SECONDARY OUTCOMES:
TCM pattern | one year
  TCM pattern is a tool for detecting the constitution among the Dry eye syndrome (DES) and healthy control.
TCM tongue diagnosis | one year
  TCM tongue diagnosis is a tool for detecting tongue expression among the Dry eye syndrome (DES) and healthy control.
Heart rate variability (HRV) | one year
  Heart rate variability (HRV) is a tool for detecting ratio betwee n High-frequency (HF) activity and low-frequency (LF) activity among the Dry eye syndrome (DES) and healthy control.
TCM pulse diagnosis | one year
  TCM tongue diagnosis is a tool for detecting tongue expression pulse pattern among the Dry eye syndrome (DES) and healthy control.
SF-36(36-Item Short Form Survey ) | one year
  SF-36 is a tool for evaluating Health-Related Quality of Life among the Dry eye syndrome (DES).
ESSPRI(EULAR Sjögren's Syndrome Patient Reported Index) | one year
  ESSPRI is a tool for evaluating the symptoms of SJS among the dry eye syndrome.
Tear breakup time (TBUT) | one year
  Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease.
Whole-genome genotyping(TWBv2.0) | one year
  By using the Whole-genome genotyping(TWBv2.0) of the immune-relate gene(RF5,TNIP1 (TNFAIP3),FCGR2B,TNF,LTA,NFKBIA,STAT4,IL-1β,IL-1R,IL-6,IL-6R,IL-8,IL-8R,IL-10,IL-10R,IL-12,IL-12R,IL-17,IL-17R,IL-18,IL-18R,IL-23,IL-23R,IL-27,IL-27R,TGF-β1,IFN-α,IFN-αR,IFN-γ,IFN-γR,TNFRSF4,BLK,CXCR5,CXCL10 to find the difference with the comparison between the dry eye syndrome and healthy control.
Oral microbiota | one year
  By using the Oral microbiota analysis to find the difference with the comparison between the dry eye syndrome and healthy control.
Blood biochemical analysis | one year
  By using the blood biochemical analysis of BUN,Cre,AST,ALT,CRP and ESR to evaluate the liver function and renal function among the Dry eye syndrome.
Cytokine biomarkers | one year
  By using cytokine biomarkers analysis of IL-17,MMP-9,BAFF and BCMA to find the difference with the comparison between the dry eye syndrome and healthy control.
CBC(complete blood count) | one year
  A complete blood count (CBC) is a blood test used to evaluate overall health among the Dry eye syndromes.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ching-Mao, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan